CLINICAL TRIAL: NCT04381546
Title: Projet GonioSEF: Etude de faisabilité d'un Dispositif d'amélioration du défaut de Report d'Appui Pendant la Marche en Phase Portante Chez Des Sujets présentant Une Atteinte du système Nerveux Central
Brief Title: FES-induced Muscular Control of the Knee on Balance and Gait Retraining After a Stroke or a Cerebral Injury
Acronym: GONIOSEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Rééducation et Réadaptation Fonctionnelle La Châtaigneraie (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-A03611-52
Record Dates: First submitted 2018-05-16; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Hemiplegia; Gait, Hemiplegic; Gait, Unsteady; Rehabilitation
MeSH Terms: conditions — Hemiplegia; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Feasibility study
Masking Description: FES-based control of knee joint to reduce stance phase asymmetry during gait in patients with post-stroke hemiplegia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FES in patients with hemiplegia (Experimental): Patients will be equipped with 5 inertial measurement units. Two wireless bluetooth pressure insoles will be connected to the Raspberry. Electrical stimulation will be delivered via a wireless stimulator to the quadriceps and hamstrings via surface electrodes. Insoles will be used to online analyze Paretic Foot Support to discriminate between stance and swing phases. Stimulation will also be delivered just before initial contact at the end of swing phase. In stance phase, stimulation will be triggered either to quadriceps or hamstrings, depending on the paretic knee angle estimation relatively to the knee angle setpoint defined by the practitioner as the optimal flexion during stance phase (around 5°).
  Interventions: Other: Functional Electrical Stimulation FES

INTERVENTIONS:
Other: Functional Electrical Stimulation FES — Functional electrical stimulation (FES) is delivered to the quadriceps and hamstrings of the paretic limb in patients with hemiplegia. It is based on the real-time estimation of the knee angle and support phase during gait.

SUMMARY:
The main hypothesis of the present study is that a safer knee joint is likely to encourage post stroke patients at an early stage to rely on their hemiparetic leg and transfer their weight onto it while walking. The main purpose of the present work is to assess the feasibility of FES-induced muscular control of the hemiplegic knee joint in order to improve stance phase support symmetry recovery in individuals with post stroke hemiplegia. Functional electrical stimulation (FES) is delivered to the quadriceps and hamstrings of the paretic limb based on the real-time estimation of the knee angle and support phase.

DETAILED DESCRIPTION:
The process of gait recovery in patients with severe post-stroke hemiplegia requires a significant investment and effort for both the patient and the therapist and is not always leading to a safe and autonomous gait. Increasing the chances for the patients of regaining a functional walking gait within limited timeframes is a challenge. Several studies have focused their attention on the neurological foot in the chronic phase because a poorly controlled foot dorsiflexion is a factor limiting gait recovery and increasing fall risk. Functional Electrical Stimulation (FES) can be used as an alternative to an orthosis to restore walking by activating paralyzed muscles. FES has been extensively studied to correct drop foot by activating foot dorsiflexors or inducing a withdrawal reflex.

Few studies have considered knee joint which has a major role, especially for the quality of the support, and this over the entire cycle of walking. In the initial phase after stroke, ensuring a safe knee control remains difficult because of the associated disorders including the lack of proprioceptive feedback. Classical observed disorders in this population are knee hyperextension during the stance phase (genu recurvatum) and flexed knees (crouch gait). Fixed orthoses are usually used to prevent this by limiting knee flexion or extension over the gait. FES is also an alternative to produce appropriately timed knee flexion or extension. Bioness L300 Plus© device proposes a thigh cuff embedding electrodes stimulating the quadriceps muscles to extend knee at the appropriate time during gait based on shank angle observation. Previous studies have investigated the contribution of quadriceps and gluteus maximus stimulation in improving standing balance and weight transfer or hamstrings stimulation associated to foot dorsiflexors stimulation in improving gait performance.

One of the main objectives of an early rehabilitation is to encourage patients with hemiplegia to rely on their paretic leg and to transfer their weight onto it while walking. Depending on the gait phase, the knee extension and flexion are restricted to a safety range by the adaptive delivery of quadriceps and hamstring electrical stimulation. A sensor network detects gait phases and knee angle evolution from which stimulation levels are modulated.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Cerebral injury or stroke
* Interval time since the onset of the neurological event: min 8 weeks (in case of an acute cerebral damage) or at a any time in case of a chronic affection
* Surface electrical stimulation of quadriceps and hamstrings possible
* Free range of motion in lower limbs
* Ankle-foot orthosis, dynamic or static
* Limited perimeter distance < 50 meters with or without walking technical aids

Exclusion Criteria:

* Knee-Ankle-Foot orthosis is required
* Body mass index > or = 30
* Thrombophlebitis
* Muscular pathology
* Unstable Cardio-Vascular pathology
* Lower limb prosthesis
* Unstable seizures
* Orthostatic hypotension
* Recent fracture in lower limbs (<12 months)
* Pacemaker
* Pregnancy
* Betablockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Assymetry of stance phase | 24 hours
  symmetry ratio of stance duration between paretic and non-paretic limbs
Assymetry of weight support in stance phase | 24 hours
  percentage of weight supported during stance phase relatively to the total weight

SECONDARY OUTCOMES:
Comfortable walking speed | 24 hours
  The preferred walking speed at which the participant choose to walk and speed at which there is least energy consumption per unit distance
Cadence | 24 hours
  The total number of full cycles on a 10m walking path
Physiological Cost Index (PCI) | 24 hours
  Energy cost in walking. PCI is the ratio of the difference in working and resting mean heart rates (bpm) and the self-selected (comfort) walking speed (m/min). The PCI value reflects the energy expenditure for walking and is expressed as heartbeats per meter.
Borg score of the exercise intensity | 24 hours
  Rating of perceived exertion while walking. Perceived effort of walking using a Borg scale from 6 (no exertion) to 20 (maximum exertion) evaluated by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Fattal, MD, PhD, Principal Investigator — Centre de Rééducation et de Réadaptation Fonctionnelle La Châtaigneraie
Locations (1):
- Centre de Rééducation et de Réadaptation Fonctionnelle La Châtaigneraie, Menucourt, France